CLINICAL TRIAL: NCT01651533
Title: Mental Practice in Chronic, Stroke-Induced Hemiparesis
Brief Title: Mental Practice in Chronic, Stroke Induced Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011H0216; NCT01026896 (obsolete NCT alias); NCT01308398 (obsolete NCT alias)
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Hemiparesis
Keywords: Mental practice group; Active control group
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Mental Practice Group (Experimental)
  Interventions: Behavioral: Mental Practice Group
- Active Comparator: Active Control Group (Active Comparator)
  Interventions: Behavioral: Active Control Group

INTERVENTIONS:
Behavioral: Mental Practice Group — Patients are administered rehabilitative therapy targeting their affected arms on 3 days/week during a ten week period. Directly after the therapy session, they participate in targeted mental practice session in which they cognitively rehearse the movement that they just physically practiced.
  Arms: Experimental: Mental Practice Group
Behavioral: Active Control Group — Individuals assigned to this group are administrated rehabilitative therapy targeting their affected arms in half four increments, occurring 3 days/week for 10 weeks. They also are administered an intervention in which they listen to a relaxation tape and/or tapes in which they receive instructions on exercises and information on stroke care.
  Arms: Active Comparator: Active Control Group

SUMMARY:
Stroke is the leading cause of disability in the United States, producing motor impairments that compromise performance of valued activities. Hemiparesis (or weakness in one arm) is particularly disabling, is the primary impairment underlying stroke-related disability, and the most frequent impairment treated by therapists in the United States. This study will test efficacy of a promising technique in reducing arm disability and increasing function, thereby improving outcomes and health, reducing care costs, for community dwelling patients with stroke-induced hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* a Fugl-Meyer score > 27, which is indicative of minimal to moderate arm impairment;
* stroke experienced > 6 months prior to study enrollment;
* minimal cognitive impairment, a score > 25 on the Folstein Mini Mental Status Examination (MMSE);
* age > 21 years old and < 80 years old;
* have experienced one clinical stroke as verified by a physician;
* discharged from all forms of physical rehabilitation targeting the affected arm.

Exclusion Criteria:

* < 21 years old;
* excessive pain in the affected hand, arm or shoulder, as measured by a score > 5 on a 10-point visual analog scale;
* excessive spasticity in the affected biceps, triceps, wrist, or fingers, as defined as a score of greater than or equal to 2 on the Modified Ashworth Spasticity Scale;
* currently participating in any experimental rehabilitation or drug studies targeting UE;
* mirrors movements(i.e., involuntary movements by the unaffected hand during attempts at unilateral movement by the stroke-affected hand during attempts at unilateral movement by the stroke-affected hand);
* history of parietal stroke (because some data suggest that ability to estimate manual motor performance through mental imagery is disturbed after parietal lobe damage);
* affected arm joint restriction that in the opinion of the investigator would hinder study participation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in movement in the affected fingers and wrist as measured by the Action Research Arm Test | 2-3 weeks before intervention; 1 week after intervention; 3 months after intervention
  This is a measure that examines the participant's ability to use the affected wrist and fingers to grasp, pinch, and grip small objects (i.e., fine motor skills). Gross movements(e.g., touching the top of the head using the affected arm) are also briefly examined. The investigator will measure changes in these abilities. We will do this by administering the measure before and after participation in the study to determine if a change occurred in patients' movement abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Page, PhD,M.S., Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Metrohealth, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio